CLINICAL TRIAL: NCT05373420
Title: COVID-19 Vaccination Uptake in Belgium: Sociodemographic and Socioeconomic Disparities - A Retrospective Cohort Study
Brief Title: COVID-19 Vaccination Uptake in Belgium : Sociodemographic and Socioeconomic Disparities
Status: Completed | Type: Observational
Sponsor: Sciensano (Other Government)
Responsible Party: Sponsor
Other Study IDs: B.U.N. 1432020000371
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccination; socioeconomic factors; sociodemographic factors; Inequity
MeSH Terms: conditions — COVID-19 | interventions — Educational Status; Sex; Health Literacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All individuals tested for COVID-19 in Belgium: All individuals of 18 years old and over tested for COVID-19 at least once in Belgium until the 31st of August 2021
  Interventions: Other: Education level; Other: Household net income; Other: Gender; Other: Migration background; Other: Household type; Other: Health literacy

INTERVENTIONS:
Other: Education level — Educational level was classified using the International Standard Classification of Education (ISCED) : ISCED0 (less than primary education), ISCED1 (primary education), ISCED2 (lower secondary school), ISCED3 (upper secondary school), ISCED4 (post-secondary non tertiary education), ISCED5 (short-cycle tertiary education), ISCED6 (bachelor's or equivalent level), ISCED7 (master's or equivalent level), ISCED8 (doctoral or equivalent level). We merged these different categories into three main education level : low (ISCED0 to ISCED2), middle (ISCED3 to ISCED4) and high (ISCED5 to ISCED 8). This information is provided by STATBEL.
Other: Household net income — Income information is available as deciles of the net income of the whole household. This indicator is further categorized into low income (deciles 1 to 4), middle income (deciles 5 to 7), and high income (deciles 8 to 10). This information is provided by STATBEL.
Other: Gender — Male or female. This variable is obtained from the Belgian national registry.
Other: Migration background — Migration background is based on the first nationality and the parents' country of origin. This variable distinguishes between native-born individuals, second-generation migrants, first-generation European migrants, and first-generation non-European migrants. This information is provided by STATBEL.
Other: Household type — Household type provides a partial picture of the social environment and is distinguished between one person, couples, couples with children, single parents, other, collectivity (prison, nursing homes, religious community, etc.). This information is provided by STATBEL.
Other: Health literacy — Having a health care degree is used as a proxy for health literacy and is provided by CoBRHA. The scientific and medical background can lead to more preventive and responsible behaviors towards infectious diseases. Moreover, being a health professional can lead to the need to protect patients and themselves against infections, without necessarily having very advanced knowledge of infectious diseases and vaccines.

SUMMARY:
In January 2021, the vaccination campaign against coronavirus disease 2019 (COVID-19) started in Belgium. The vaccination campaign was conducted in several phases, with the first phase targeting priority groups starting in January 2021. The second phase began in June 2021 with the invitation of everyone aged 18 years and older before extending access to 12 years and older from summer 2021. Children aged 5-11 were also invited for vaccination from December 2021 onwards.

The presence of a social gradient in COVID-19 infections and subsequent outcomes has been clearly demonstrated. Individuals from lower socioeconomic groups, for example with lower income, lower education level or unemployed are more likely to be infected by the SARS-CoV-2 and to develop severe complications after the infection such as hospitalization, ICU admission or death. Certain sociodemographic characteristics such as male gender, older age, living in crowded households, or belonging to ethnic/racial minorities are also associated with a higher risk of COVID-19 infection and severe outcomes. In addition to disparities in infection, hospitalization and mortality, some studies have also documented a lower COVID-19 vaccination coverage among people from disadvantaged socioeconomic groups during COVID-19 pandemic.

Despite widespread vaccine promotion efforts and the fact that Belgium has the 7th highest full vaccine coverage in the European Union (89% of people over 18 years old had completed their primary course of vaccination on 08 April 2022), concerns regarding vaccine equity remain. Vaccine uptake depends on a range of factors, including the socio-cultural environment, pre-existing health needs and individual choice. Identifying differences in vaccination between population groups is crucial to assess the effectiveness of the vaccination strategy in Belgium and its relationship to the further spread of COVID-19.

The objective is to identify whether vaccination coverage has been equitable across Belgium and, if not, which groups of individuals are less likely to be covered by the COVID-19 vaccine, with respect to their sociodemographic (SD) and socioeconomic (SE) characteristics.

This study therefore aims to highlight SD and SE disparities in the uptake of the first dose of COVID-19 vaccine in Belgium among people of 18 years and over.

DETAILED DESCRIPTION:
1. Study design and data sources

   In this retrospective cohort study, the investigators aimed to unravel SE and SD disparities in the uptake of the first COVID-19 vaccine dose using data from the LINK-VACC project. This project was launched by Sciensano, the institute legally responsible for the surveillance of infectious diseases in Belgium (Royal Decree of 21/03/2018), to perform the post-authorization surveillance of COVID-19 vaccines in Belgium.

   To that aim, selected variables from multiple existing national health and social sector registries were linked at an individual level using the unique Belgian social security number. The databases were linked within a pseudonymised environment hosted by Healthdata.be of Sciensano. For the present study, four databases were used :
   * Vaccinnet+, the Belgian vaccine registry, which contains information on all COVID-19 vaccine doses administrated in Belgium. It includes demographical data of the vaccinated person (sex, age, postal code of residence), as well as data on the vaccinator (type (person or organization) and postal code) and on the administrated vaccine (brand of the vaccine, lot number, date of administration, date of registration).
   * The COVID-19 Healthdata database containing data from COVID-19 laboratory tests performed in Belgium (data of sampling and test result).
   * The STATBEL database provided by the Belgian Statistical Institute which contains variables related to socioeconomic and sociodemographic characteristics.
   * The Common Base Registry for HealthCare Actor (CoBRHA) allowing the identification (by profession and specialty) of people who have been licensed to practice a healthcare profession in Belgium.
2. Cohort definition

   The population of interest includes all individuals of 18 years and older tested for COVID-19 at least once in Belgium until the 31st of August 2021 (which is the date of linkage between STATBEL, Vaccinnet+ and the COVID-19 Healthdata database) for whom SD and SE information from STATBEL database was available.

   The cohort is built from Vaccinnet+ and the COVID-19 Healthdata database which includes all doses of vaccines administered and PCR and rapid antigenic tests performed in Belgium, respectively. As of 31 August 2021, 10 475 908 individuals had been tested and/or vaccinated at least once in Belgium according to Vaccinnet+ and the COVID-19 Healthdata database. On January 1, 2021, the official Belgian population included 11 521 238 inhabitants, demonstrating a high coverage of the total Belgian population by these two data sources (90.92%).

   The relevant SE and SD variables were then included after linking with STATBEL database based on the individual national identification number. The data source available from STATBEL contains SE and SD information for 10 309 300/10 475 908 individuals registered at least once either in Vaccinnet+ from 28 December 2020 to 31 August 2021 or in the COVID-19 Healthdata database before 31 August 2021, corresponding to a linkage rate of 98.41%. Information on the healthcare license available in CoBRHA were then added. After these linkages, people who were deregistered, migrated and deceased based on their status in the national registry were excluded. People whose age, region or gender were unknown were also excluded.

   In order to be able to compare vaccination rate according to each SE and SD indicators, the investigators included only individuals tested before 31 August 2021 since it is the date of linkage between Vaccinnet+, COVID-19 Healthdata database and STATBEL. Finally, individuals under 18 years of age were excluded as they were considered as a group in their own right in the vaccination strategy by being vaccinated the latest in a separate phase of the vaccination campaign.

   The final cohort for this study is therefore composed of 5 341 584 individuals of 18 years and over tested in Belgium until the 31st of August 2021.
3. Outcome The outcome variable, provided by Vaccinnet+, is the uptake of the first dose of COVID-19 vaccine until the 31st of August 2021. The investigators considered that, at this date, all individuals over 18 years of age had received an invitation to be vaccinated with the first dose and had the opportunity to receive this dose of vaccine in Belgium.

ELIGIBILITY:
Inclusion criteria :

* Tested at least once in Belgium before 31 August 2021

Exclusion criteria :

* people with a national registry status equivalent to deceased
* people with a national registry status equivalent to migrated
* people with a national registry status equivalent to deregistered
* people with an unknown age
* people with an unknown gender
* people with an unknown region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals of 18 years and over tested for COVID-19 at least once in Belgium before 31 August 2021
Sampling Method: Non-Probability Sample
Enrollment: 5341584 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who received the first dose of COVID-19 vaccine | 28 December 2020 - 31 August 2021
  Uptake of the first COVID-19 vaccine dose until the 31st of August 2021 in Belgium

CONTACTS AND LOCATIONS:
Overall Officials: Lucy LC Catteau, PhD, Principal Investigator — Sciensano
Locations (1):
- Lisa Cavillot, Brussels, Belgium

REFERENCES:
- See also: Vaccination | Coronavirus COVID-19 — http://www.info-coronavirus.be/fr/vaccination/
- See also: COUVERTURE VACCINALE ET IMPACT ÉPIDÉMIOLOGIQUE DE LA CAMPAGNE DE VACCINATION COVID-19 EN BELGIQUE — https://covid-19.sciensano.be/sites/default/files/Covid19/COVID-19_THEMATIC_REPORT_VaccineCoverageAndImpactReport_FR.pdf
- See also: Association of race, ethnicity, and community-level factors with COVID-19 cases and deaths across U.S. counties — http://pubmed.ncbi.nlm.nih.gov/33285500/
- See also: Community-Level Factors Associated With Racial And Ethnic Disparities In COVID-19 Rates In Massachusetts — https://pubmed.ncbi.nlm.nih.gov/32853056/
- See also: Social Determinants of COVID-19 in Massachusetts, United States: An Ecological Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7411251/
- See also: Derivation and Validation of Clinical Prediction Rules for COVID-19 Mortality in Ontario, Canada — https://pubmed.ncbi.nlm.nih.gov/33204755/
- See also: COVID-19 clinical outcomes and nationality: results from a Nationwide registry in Kuwait — https://bmcpublichealth.biomedcentral.com/articles/10.1186/s12889-020-09490-y
- See also: Factors Associated With Racial Differences in Deaths Among Nursing Home Residents With COVID-19 Infection in the US — https://pubmed.ncbi.nlm.nih.gov/33566110/
- See also: COVID-19 fatality in Mexico's indigenous populations — https://pubmed.ncbi.nlm.nih.gov/33743216/
- See also: Variation in racial/ethnic disparities in COVID-19 mortality by age in the United States: A cross-sectional study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7575091/
- See also: Ethnic-minority groups in England and Wales-factors associated with the size and timing of elevated COVID-19 mortality: a retrospective cohort study linking census and death records — https://pubmed.ncbi.nlm.nih.gov/33349855/
- See also: Laboratories | Database COVID-19 TestResults — https://covid19lab.healthdata.be/data-providers/laboratories
- See also: Are we really all in this together? The social patterning of mortality during the first wave of the COVID-19 pandemic in Belgium — https://researchportal.vub.be/en/publications/are-we-really-all-in-this-together-the-social-patterning-of-morta
- See also: The income gradient in mortality during the COVID-19 crisis: evidence from Belgium — http://www.andredecoster.be/publication/the-income-gradient-in-mortality-during-the-covid-19-crisis-evidence-from-belgium-2/
- See also: COVID-19 BULLETIN EPIDEMIOLOGIQUE HEBDOMADAIRE — https://covid-19.sciensano.be/sites/default/files/Covid19/COVID-19_Weekly_report_FR.pdf
- See also: Health literacy and infectious diseases: why does it matter? — https://pubmed.ncbi.nlm.nih.gov/26751238/
- See also: Attitudes of healthcare workers towards COVID-19 vaccination: a survey in France and French-speaking parts of Belgium and Canada, 2020 — https://pubmed.ncbi.nlm.nih.gov/33478623/
- See also: COVID-19 Vaccine Acceptance among Health Care Workers in the United States — https://pubmed.ncbi.nlm.nih.gov/33546165/
- See also: COVID-19 Vaccination Acceptance Among Healthcare Workers and Non-healthcare Workers in China: A Survey. Frontiers in Public Health — https://www.frontiersin.org/article/10.3389/fpubh.2021.709056
- See also: Conceptual causal framework to assess the effect of SARS-CoV-2 variants on COVID-19 disease severity among hospitalized patients — https://www.sciensano.be/en/biblio/conceptual-causal-framework-assess-effect-sars-cov-2-variants-covid-19-disease-severity-among
- See also: Structure de la population — https://statbel.fgov.be/fr/themes/population/structure-de-la-population#panel-13
- See also: Weekly report-Sciensano — https://www.phrasebank.manchester.ac.uk/introducing-work/